CLINICAL TRIAL: NCT00541151
Title: Long-Term Effectiveness Trial for AMS Sling Systems
Brief Title: MiniArc Study: Long-Term Effectiveness Trial for AMS Sling Systems
Acronym: MiniArc
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: American Medical Systems (Industry)
Responsible Party: Audrey Singh- Clinical Project Lead, American Medical Systems, Inc.
Other Study IDs: WC0605
Record Dates: First submitted 2007-10-05; First posted 2007-10-10 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2010-08

CONDITIONS: Stress Urinary Incontinence in Women
Keywords: Stress urinary incontinence in Women

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: MiniArc — sling system
  Other Names: MiniArc or single incision sling

SUMMARY:
Multi-center, prospective, single arm study. Qualify patients will receive treatment for stress urinary incontinence by implantation of an AMS Sling System. The study is a long-term evaluation of effectiveness and safety associated with AMS sling systems.

DETAILED DESCRIPTION:
This study is a post market study to evaluate variables of the implantation, safety, and outcomes in a representative population (SUI) indicated for AMS sling systems at various time points. The study duration is 2 year with an estimated 200 enrollment. The outcomes of the treatment will be evaluated via pad weight test, cough stress test, QoLs,and other patient administered questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Females 18 years or older who have confirmed SUI defined as involuntary loss of urine that occurs during physical activity, such as coughing, sneezing, laughing, or exercise.

Exclusion Criteria:

* Unwilling or unable to sign ICF
* Unable to understand the study or has a history of non-compliance with medical devices
* Contradicted for the implantation surgery due to the following: renal sufficiency, urethral diverticulum, fistula, significant prolapse conditions, pregnant, pelvic cancer, compromise immune system,vulvar pain,blood coagulation disorder, and chronic abscesses
* Pelvic prolapse greater than grade 3
* Is, in the investigator's opinion, otherwise unsuitable for the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Females 18 years or older who have confirmed SUI
Sampling Method: Non-Probability Sample
Enrollment: 188 (Actual)
Dates: Start 2007-09; Primary Completion 2010-08 (Estimated); Study Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
Evaluation of long-term effectiveness after implantation of MiniArc sling via qualitative(i.e.UDI-6 and IIQ-7) and quantitative measurement (i.e.pad weight test and cough stress test) in females for treatment of SUI in general post-market use. | 2 years

SECONDARY OUTCOMES:
Evaluation of procedural variables of the implantation,outcomes,and long-term safety.These outcomes will be measured via questionnaires, procedural data, and report of adverse events. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kennelly, MD, Principal Investigator — McKay Urology Research
Locations (1):
- McKay Urology Research, Charlotte, North Carolina, United States